CLINICAL TRIAL: NCT05623527
Title: Clinical Characteristics and Prognosis of Acute Cerebrovascular Events Secondary to Patients Receiving Cardiac Electronic Implants (SOS-CARE) - A Multicenter Real-world Trial
Brief Title: Clinical Characteristics and Prognosis of Acute Cerebrovascular Events Secondary to Patients Receiving Cardiac Electronic Implants
Acronym: SOS-CARE
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2022LSK-408
Record Dates: First submitted 2022-10-27; First posted 2022-11-21 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2023-10

CONDITIONS: Stroke; Atrial Fibrillation; Pacemaker
MeSH Terms: conditions — Stroke; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ischemic stroke group: 1. Ischemic stroke secondary to patients receiving cardiac electronic implants
  2. Ischemic stroke met the diagnostic criteria of the 2018 edition of the Chinese Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke, and was confirmed by cranial CT/MRI scan.
  Interventions: Device: cardiac electronic implants
- Transient ischemic attack group: 1. Transient ischemic attack secondary to patients receiving cardiac electronic implants
  2. Ischemic stroke met the diagnostic criteria of the 2018 edition of the Chinese Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke, and was confirmed negative of new onset of infarction by cranial CT/MRI scan.
  Interventions: Device: cardiac electronic implants
- Cerebral hemorrhage group: 1. Cerebral hemorrhage secondary to patients receiving cardiac electronic implants
  2. Cerebral hemorrhage met the diagnostic criteria of the 2021 Chinese Guidelines for the Diagnosis and Treatment of cerebral hemorrhage and was confirmed by head CT/MRI.
  Interventions: Device: cardiac electronic implants

INTERVENTIONS:
Device: cardiac electronic implants — Cardiac electronic implants(CIED) includes permanent pacemaker (PPM), implantable cardioverter defibrillator (ICD), three-chamber pacemaker for cardiac resynchronization therapy defibrillator, lead free pacemaker, etc.

SUMMARY:
To investigate the incidence, clinical characteristics and prognosis of acute ischemic and hemorrhagic cerebrovascular disease secondary to the implantation of cardiovascular implantable electronic devices, so as to provide a basis for subsequent treatment strategies and risk factor stratification.

This study intends to retrospectively collect the incidence and case characteristics of acute cerebral infarction, cerebral embolism, transient ischemic attack and cerebral hemorrhage in CIED patients admitted to the First Affiliated Hospital of Xi 'an Jiaotong University and other centers from January 2012 to September 2022. Then, the incidence of poor prognosis and related factors of patients within 3 months were followed up by telephone to provide a basis for subsequent treatment strategy and risk factor stratification.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute cerebrovascular disease secondary to cardiac electronic device implantation.
* Hospitalized from January 2012 to September 2022.

Exclusion Criteria:

* Patients were absent of cranial CT/MRI scan data.
* Patients refuse to take follow-up interviews.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From January 2012 to September 2022, any patients with cardiac implantable electronic device
Sampling Method: Probability Sample
Enrollment: 13324 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
The incidence of acute cerebrovascular disease | About 4 weeks after the enrollment
  Number and rate of patients with acute cerebrovascular disease secondary to patients receiving cardiac electronic implants. The data were obtained from the medical records.

SECONDARY OUTCOMES:
In-hospital mortality | About 4 weeks after the enrollment
  In-hospital mortality of acute cerebrovascular disease in patients receiving cardiac electronic implants. The data were obtained from the medical records.
All-cause mortality | 3 months after the enrollment
  All-cause mortality within 3 months of telephone follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Guoliang Li, Principal Investigator — Xi'an Jiaotong University First Affiliated Hospital
Locations (1):
- Guoliang Li, Xi'an, Shannxi Province, China

IPD SHARING:
Plan to Share IPD: Undecided